CLINICAL TRIAL: NCT05379790
Title: Concomitant Intraperitoneal and Systemic Chemotherapy in Patients With Extensive Peritoneal Carcinomatosis of Gastric Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. R.H.J. Mathijssen, MD, PhD, Principal Investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL79619.078.21
Record Dates: First submitted 2022-04-25; First posted 2022-05-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer; Peritoneal Metastases
Keywords: Peritoneal metastases; Gastric cancer; Intraperitoneal; Irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: A classic phase I '3+3' dose-escalation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Intraperitoneal irinotecan 50 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 1 50 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX
- Intraperitoneal irinotecan 75 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 2 75 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX
- Intraperitoneal irinotecan 100 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 3 100 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX
- Intraperitoneal irinotecan 150 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 4 150 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX
- Intraperitoneal irinotecan 200 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 5 200 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX
- Intraperitoneal irinotecan 250 mg + CAPOX (Experimental): Intraperitoneal irinotecan, dose level 6 250 mg flat dose + oral capecitabine and systemic oxaliplatin (CAPOX) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: CAPOX

INTERVENTIONS:
Drug: Irinotecan — 3 weekly IP irinotecan (max 6 cycles), dose via dose-escalation design as specified per arm.
  Other Names: Intraperitoneal irinotecan
Drug: CAPOX — Capecitabine 1000 mg/m2 twice daily day 1-14 (per os), and Oxaliplatin 130 mg/m2 on day 1 IV infusion.

SUMMARY:
Gastric cancer with peritoneal carcinomatosis has a poor prognosis, with little treatment options available. The current treatment strategy consists of palliative systemic chemotherapy. However, previous research suggests that systemic chemotherapy is less effective against peritoneal carcinomatosis than against metastases that spread hematogenously.

Several studies suggested that in patients with peritoneal carcinomatosis, intraperitoneal chemotherapy (IP) may be superior compared to intravenous chemotherapy. Intraperitoneal chemotherapy could lead to higher concentrations of chemotherapy in the peritoneal cavity for a longer period of time, resulting in an increased cumulative exposure to the peritoneal metastases. A few Asian studies have shown promising results with intraperitoneal chemotherapy in patients with peritoneal carcinomatosis of gastric origin. However, intraperitoneal chemotherapy combined with systemic chemotherapy has not been investigated in Western patients with peritoneal carcinomatosis of gastric origin yet. The objective of this trial is to establish the maximum tolerated dose (MTD) of intraperitoneal administration of irinotecan, added to systemic capecitabine/oxaliplatin (CAPOX) in patients with peritoneal carcinomatosis of gastric origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of HER2-negative gastric cancer.
* A histologically confirmed diagnosis of peritoneal carcinomatosis.
* Age ≥ 18 years old.
* Written informed consent according to the ICH-GCP and national/local regulations.
* A peritoneal cancer index (PCI) ≥7 evaluated by laparoscopy or laparotomy before inclusion in this trial.
* Patients must be ambulatory: World Health Organisation (WHO) performance status 0 or 1.
* Life expectancy of at least 3 months.
* Ability to return to the Erasmus MC for adequate follow-up as required by this protocol.
* Patients must have normal organ function and adequate bone marrow reserve as assessed by the following laboratory requirements:

  * absolute neutrophil count >1.5 * 10^9/l;
  * platelet count >100*10^9/l;
  * Hb>6.0mmol/l;
  * Bilirubin < 1.5x upper limit of normal (ULN);
  * Serum aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2.5 x ULN;
  * Glomerular Filtration Rate (GFR) >45 and Creatinine clearance <2 x ULN.

Exclusion Criteria:

* Medical or psychological impediment to probable compliance with the protocol.
* Serious concomitant disease or active infections.
* Distant metastasis other than peritoneal metastasis or metastatic lymph nodes.
* No sufficient oral food intake.
* Polyneuropathy grade 2 or worse according to CTCAE version 5.0.
* History of auto-immune disease or organ allografts, or with active or chronic infection, including HIV and viral hepatitis.
* Serious intercurrent chronic or acute illness such as pulmonary (COPD or asthma) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for participation in this study.
* Homozygous UGT1A1*28 genotype.
* Homozygous dihydropyrimidine dehydrogenase (DPYD) genotype (tested for *2A, *13, 2846A>T, and 1236G>A).
* Current use of strong CYP3A4-inhibitors or inducers. If patients use this CYP3A4-modulating medication, it is allowed to stop it within 14 days of start of treatment.
* Pregnant or lactating women.
* Concomitant participation in a competing clinical study.
* Absence of assurance of compliance with the protocol.
* An organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent, and preclude participation in the full protocol and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose | 18 weeks
  The maximum tolerable dose and recommended phase II dose of intraperitoneal irinotecan added to systemic chemotherapy (capecitabine/oxaliplatin)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 18 weeks
  Toxicity graded according to the CTCAE v.5.0 determined at every cycle by the medical oncologist. Toxicity will be summarized descriptively.
Area Under the Curve (AUC) ratio intraperitoneal/systemic irinotecan | 3 weeks
  During the first irinotecan intraperitoneal cycle, pharmacokinetic measurements wil be obtained. These will be withdrawn at specific time-points, namely prior to infusion, at the end of the intraperitoneal infusion, ass well as 30 minutes, 1, 1.5, 2, 3, 4, 6, and 24 hours post infusion. Blood samples from a peripheral venous catheter and peritoneal fluid will be drawn from the peritoneal access port. We assume that the AUC of irinotecan and SN-38 follow a log-normal distribution. Therefore, the analysis will be performed on log-transformed data. The antilog will be taken from the ratio and corresponding 95% confidence interval boundaries will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Mathijssen, Professor, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Catharina Hospital, Eindhoven

IPD SHARING:
Plan to Share IPD: No